CLINICAL TRIAL: NCT03638232
Title: Myeloma Treatment in Real Life : Pharmacoepidemiological Approach in Midi-pyrénées
Brief Title: Myeloma Treatment in Real Life
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: 14 7439 07
Record Dates: First submitted 2018-08-16; First posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Multiple Myeloma
Keywords: Drug consumption; Response to treatment; Non optimal drug use
MeSH Terms: conditions — Multiple Myeloma | interventions — Routinely Collected Health Data; Electronic Health Records

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with multiple myeloma: Data to be collected are :
  * Drug exposition data
  * Administrative data
  * Medical data
  Interventions: Other: Administrative data; Other: Medical data; Other: Drug exposition data

INTERVENTIONS:
Other: Administrative data — Gender Birthdate Department and town of residence Date of death Affiliation to french Universal Health Coverage
Other: Medical data — Long term affection code, number and medical codification Date of onset and end of care Codification of medical acts and consultation (With common classification of medical acts)
Other: Drug exposition data — Speciality of prescribing physician CIP code of drug Name of speciality prescribed Date of deliverance Date of prescription Number of treatment box delivered

SUMMARY:
As part of an oral treatment regimen in ambulatory practice, certain uses in connection with drug consumption associated could alter treatment outcomes observed in randomized clinical trials.

The increase in progression-free survival in myeloma may be accompanied by an impaired quality of life and a resurgence of pain symptoms over time, which could potentially lead to medication overuse involving painkillers but also psychotropic drugs. These combined consumption may affect survival through mechanisms of pharmacological or non-pharmacological interactions.

As part of this project, we wish to explore the scheme of adherence to myeloma drugs, and thus validate the decision diagram of hypothesis of not adequate of drug use in ambulatory conditions, from observational data. This discrepancy could result from poor adherence or suboptimal drug use but also from concomitant exposures to other drugs which may interact with myeloma. Before considering a study of greater magnitude that could address the consequences of non optimal drug use on clinical response criteria, such as duration of response or survival, it seems appropriate to confirm these assumptions within ' an exploratory study.

ELIGIBILITY:
Inclusion Criteria:

* Beneficiaries or entitled to health insurance or covered by the national system of information of health insurance
* Identified as multiple myeloma
* Incident patient : Subject presenting none of inclusion criteria during the 6 months observation period

Exclusion Criteria:

* Non incident patient : Subject presenting at least one of inclusion criteria during the 6 months observation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with multiple myeloma in Midi-Pyrénées
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of myeloma treatment observance in real life as assessed by data collected in french national system of information of health insurance | Through the end of study (15 months)

SECONDARY OUTCOMES:
Description deliverance scheme of treatment used in multiple myeloma as assessed by data collected in french national system of information of health insurance | Through the end of study (15 months)
Evaluation of respect of official recommendation related to observance in multiple myeloma treatment as assessed by expression of Medication Possession Ratio (MPR) | Through the end of study (15 months)
  The Medication Possession Ratio (MPR) measure compliance of prescriber with official recommendations and the one for the patient in relation to the prescription by evaluating the difference between the quantities delivered and the theoretical quantities calculated in joining recommended intake scheme. It is estimated by the ratio of number of defined daily doses delivered over a given period and the number of theoretical defined daily doses if maximum observance
Description of care consumption in multiple myeloma as assessed by data collected in french national system of information of health insurance | Through the end of study (15 months)

CONTACTS AND LOCATIONS:
Overall Officials: Lapeyre-Mestre Maryse, PHD, Study Director — University Hospital of Toulouse

IPD SHARING:
Plan to Share IPD: No